CLINICAL TRIAL: NCT02163772
Title: Early Intracordal Hyaluronic Acid Injection During Spontaneous Reinnervation for Unilateral Recurrent Laryngeal Nerve Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSC100-2314-B-182-021
Record Dates: First submitted 2014-06-10; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2013-07

CONDITIONS: Paralysis, Unilateral, Vocal Cord
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intracordal hyaluronate injection (HI) (Experimental): The intervention of Intracordal hyaluronate (Restylane) injection is given in this group No other therapies are given
  Interventions: Procedure: Intracordal hyaluronate injection
- Conservative management (CM) (No Intervention): In this arm, only observation is arranged. No therapy is given.

INTERVENTIONS:
Procedure: Intracordal hyaluronate injection
  Other Names: Resylane
  Arms: Intracordal hyaluronate injection (HI)

SUMMARY:
Backgrounds: Unilateral vocal cord paralysis caused from recurrent laryngeal nerve (RLN) injury is not an unusual disease and may deteriorate patients'voice and swallowing outcomes. Although the long term treatment effect is encouraged, the point when to perform surgical treatment is not conclusive. Previous reports suggested late treatment principle because patients may spontaneous reinnervation to some degree within 4-5 months after injury. The vocal cord position and tone may change during reinnervation. Others delineated laryngeal synkinesis by misdirected reinnervation is common and suggested early temporary injection laryngoplasty. They implied early injection laryngoplasty may improve patients'not only short term voice outcomes but also decrease the incidence of transcervical laryngeal framework surgery as a determined surgery. However, lacking of prospective study and objective data makes the treatment-time policy still controversial. Purposes: 1. To find incidence of spontaneous reinnervation or synkinetic regeneration. 2. To detect the relationship between changing of glottal gap and laryngeal synkinesis. 3. To detect the impaction of early intracordal hyaluronic acid injection on vocal cord position change in patients with laryngeal synkinesis. Study design: Forty patients is planned to be enrolled in the study. Twenty of them will undergo hyaluronate intracordal injection at three-six month from RLN damage. The other 20 patients will follow the watch-and wait policy. Laryngoscope, laryngeal EMG (electromyography), voice analysis and voice outcome survey will be done at 3-6 month and 12-month after RLN injury. At the end of follow up, the glottal gap, voice laboratory data and quality of life will be compared. The outcomes will also be correlated with laryngeal electromyography (LEMG) data and the impact of synkinetic reinnervation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of untreated unilateral vocal cord paralysis with a known cause of RLN injury within 3-6 month will be enrolled

Exclusion Criteria:

* Patients proved to be not suitable for transcutaneous intracordal injection under topical anesthesia. Those who had previous phonosurgery or can't follow the observation rule will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
voice outcome | before intervention and at 6 month follow-up
  VOS score: The VOS originally developed by Gliklich et al. comprises a five-item survey that evaluates the physical and social problems associated with unilateral vocal fold palsy.

SECONDARY OUTCOMES:
laryngeal electromyography | before and 6 months post intervention
  laryngeal electromyography signals were obtained using a concentric needle electrode with the surface-ground electrode adhered to the forehead. We examined the electromyography signals on bilateral thyroarytenoid muscle and cricothyroid muscles. With the concentric needle electrode in the thyroarytenoid muscle , the patient was asked to produce three series of "e"s at three different intensities (low, moderate and highest possible), with each "e" lasting at least 400 ms and each inter-"e" interval lasting about 200 ms. To evaluate cricothyroid function, the patients were asked to produce a glissando upward "e" at normal loudness.
videolaryngostroboscopy | before and 6 months post intervention
  An image of glottis was captured during the videolaryngoscopy examination while the patient vocalized /eee/ at modal pitch and regular loudness. The images showing the narrowest vocal slitglottal gap from several phonatory cycles were measured.
laboratory voice analysis | before and 6 months post intervention
  In a sound-insulated room, the patient read a standard passage and a sustained vowel at a conversational pitch and loudness. The patient's voice was captured using a unidirectional dynamic microphone (Shure SM48; Shure Brothers Inc., Agua Prieta, Mexico).
health related quality of life (SF-36) | before and 6 months post intervention
  The SF-36 questionnaire is designed for general health measurement of 8 domains, including physical functioning, role functioning-physical problems, bodily pain, general health, vitality, social functioning, role functioning-emotional problems, and mental health. The recall period of SF-36 is 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

REFERENCES:
- [Derived] Pei YC, Fang TJ, Hsin LJ, Li HY, Wong AM. Early hyaluronate injection improves quality of life but not neural recovery in unilateral vocal fold paralysis: an open-label randomized controlled study. Restor Neurol Neurosci. 2015;33(2):121-30. doi: 10.3233/RNN-140439. PMID 25588457